CLINICAL TRIAL: NCT00542009
Title: A 12-Week, Phase 2A, Randomized, Subject And Investigator Blinded, Placebo-Controlled Trial To Evaluate The Safety, Tolerability And Efficacy Of CE-326,597 On Glucose Control And Body Weight In Overweight Adult Subjects With Type 2 Diabetes Mellitus
Brief Title: A Trial In Diabetic Patients To Assess Effect Of CE-326,597 On Glucose Control And Body Weight
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A7211005
Record Dates: First submitted 2007-10-05; First posted 2007-10-10 (Estimated); Last update posted 2012-11-07 (Estimated); Status verified 2012-11

CONDITIONS: Weight Management; Treatment Of Obesity
Keywords: Phase 2A, safety and efficacy trial with CE-326,597 in patients with T2DM.

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- CE-326,597 100 mg QD (Experimental)
  Interventions: Drug: CE-326,597 100 mg QD
- CE-326,597 50 mg QD (Experimental)
  Interventions: Drug: CE-326,597 50 mg QD
- CE-326,597 25 mg QD (Experimental)
  Interventions: Drug: CE-326,597 25 mg QD
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- CE-326,597 5mg QD (Experimental)
  Interventions: Drug: CE-326,597 5mg QD

INTERVENTIONS:
Drug: CE-326,597 100 mg QD — Administered orally, once daily with morning meal for duration of trial (84 days).
  Arms: CE-326,597 100 mg QD
Drug: CE-326,597 50 mg QD — Administered orally, once daily with morning meal for duration of trial (84 days).
  Arms: CE-326,597 50 mg QD
Drug: CE-326,597 25 mg QD — Administered orally, once daily with morning meal for duration of trial (84 days).
  Arms: CE-326,597 25 mg QD
Drug: Placebo — Placebo to match CE-326,597 tablets to be administered orally, once daily with morning meal for duration of trial (84 days).
  Arms: Placebo
Drug: CE-326,597 5mg QD — Administered orally, once daily with morning meal for duration of trial (84 days).
  Arms: CE-326,597 5mg QD

SUMMARY:
Study of whether the investigational drug CE-326,597 improves glucose control and results in body weight loss in patients with type 2 diabetes

ELIGIBILITY:
Inclusion Criteria:

Patients with type 2 diabetes, not on any or on oral (up to 2) anti-diabetic medications, otherwise medically stable.

Exclusion Criteria:

Women of childbearing potential, people with unstable medical conditions, people with gallstones

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2007-12; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Glucose control | At Day 84
Body weight | At Day 84

SECONDARY OUTCOMES:
Regimen (dose or number) of anti-diabetic agents | At Day 84
GlycoMark | On Day 84
Waist circumference | On Day 84
Proportion of subjects who achieve HbA1C <7% and <6.5% | On Day 84
Population PK to analyze CE-326,597 concentrations as well as explore relationship of concentration to effect on HbA1C and body weight over duration of trial. | Throughout Study
Standard safety (via AEs, SAEs, vitals, 12-lead ECG, abdominal ultrasound) will be monitored throughout the trial. | Throughout Study
Change in following parameters: Post-prandial and fasting glucose, and insulin | On Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (48):
- United States (26):
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Fresno, California
  - Pfizer Investigational Site, National City, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Ocala, Florida
  - Pfizer Investigational Site, West Palm Beach, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Conyers, Georgia
  - Pfizer Investigational Site, Honolulu, Hawaii
  - Pfizer Investigational Site, Idaho Falls, Idaho
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Overland Park, Kansas
  - Pfizer Investigational Site, Bethesda, Maryland
  - Pfizer Investigational Site, Chaska, Minnesota
  - Pfizer Investigational Site, Minneapolis, Minnesota
  - Pfizer Investigational Site, Jackson, Mississippi
  - Pfizer Investigational Site, Henderson, Nevada
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, Fargo, North Dakota
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Lansdale, Pennsylvania
  - Pfizer Investigational Site, Rapid City, South Dakota
  - Pfizer Investigational Site, Beaumont, Texas
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Richmond, Virginia
- Bulgaria (3):
  - Pfizer Investigational Site, Pleven
  - Pfizer Investigational Site, Sofia
  - Pfizer Investigational Site, Stara Zagora
- Canada (5):
  - Pfizer Investigational Site, Coquitlam, British Columbia
  - Pfizer Investigational Site, Winnipeg, Manitoba
  - Pfizer Investigational Site, London, Ontario
  - Pfizer Investigational Site, Laval, Quebec
  - Pfizer Investigational Site, Montreal, Quebec
- India (4):
  - Pfizer Investigational Site, Bangalore, Karnataka
  - Pfizer Investigational Site, Indore, Madhya Pradesh
  - Pfizer Investigational Site, Nagpur, Maharashtra
  - Pfizer Investigational Site, Nashik, Maharashtra
- Mexico (3):
  - Pfizer Investigational Site, Ladrón de Guevara, Guadalajara, Jalisco
  - Pfizer Investigational Site, Guadalajara, Jalisco
  - Pfizer Investigational Site, Monterrey, Nuevo León
- Puerto Rico (3):
  - Pfizer Investigational Site, Ponce
  - Pfizer Investigational Site, San Juan
  - Pfizer Investigational Site, Tao Baja
- Spain (4):
  - Pfizer Investigational Site, Barcelona, Barcelona
  - Pfizer Investigational Site, Santiago de Compostela, La Coruña
  - Pfizer Investigational Site, Madrid, Madrid
  - Pfizer Investigational Site, Seville, Sevilla

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A7211005&StudyName=A%20Trial%20In%20Diabetic%20Patients%20To%20Assess%20Effect%20Of%20CE-326%2C597%20On%20Glucose%20Control%20And%20Body%20Weight